CLINICAL TRIAL: NCT00382317
Title: A Clinical Study of Iobitridol in Multislice CT Abdominal Angiography Indications
Brief Title: A Clinical Study of Iobitridol in Patients Undergoing Multislice Computed Tomography (CT) Abdominal Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ISO-44-009
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-11

CONDITIONS: Diagnostic Imaging
Keywords: MSCT indications
MeSH Terms: interventions — iobitridol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Iobitridol

SUMMARY:
This is a clinical study of iobitridol in patients undergoing multislice CT (MSCT) abdominal angiography.

ELIGIBILITY:
Inclusion Criteria:

* Male or female having reached legal majority age and up to 85 years included.
* Scheduled for an aorta and abdominal arterial tree evaluation by MSCT, either for pre-therapeutic evaluation or for post-surgical control or follow-up (including patients with prosthetic vascular material).
* Female of childbearing potential must have effective contraception (contraceptive pill or intra-uterine device), or be surgically sterilised, or post-menopausal (minimum 12 months amenorrhea) or must have a documented negative urine and/or blood pregnancy test at screening.

Exclusion Criteria:

* Patients with overt non-compensated heart failure.
* Patients with hemodynamic instability.
* Patients with ESC (European Society of Cardiology)/ESH (European Society of Hypertension) grade 3 hypertension (SBP [systolic blood pressure) over or equal to 180 mm Hg or DBP [diastolic blood pressure] over or equal to 110 mm Hg)
* Patients with known severe renal failure (defined as creatinine clearance < 30 ml/min as calculated by the Cockroft and Gault formula).
* Patients who have received diuretic or biguanide treatment during the 48 hours preceding the MSCT scan.
* Patients with known thyreotoxicosis.
* Patients with history of immediate or delayed major hypersensitivity reaction to iodinated contrast media.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Dubourdieu, PhD, Study Chair — Guerbet
Locations (2):
- AKH, Vienna, Austria
- CHU Charles Nicolle, Rouen, France